CLINICAL TRIAL: NCT05844774
Title: The Clinical Effects of Perioperative Use of the Hypotension Prediction Index
Brief Title: Post Anaesthesia Care Hypotension Prevention
Acronym: PACH-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL81361.091
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Hypotension During Surgery
Keywords: Laparotomy; Hypotension; Goal Directed Therapy; Post-operative; Prediction; Artificial intelligence
MeSH Terms: conditions — Hypotension | interventions — Health Records, Personal

STUDY DESIGN:
Intervention Model Description: 1 control group, 1 intervention group without cross-over
Masking Description: Open label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPI-intervention algorithm (Experimental): In the intervention group the HemoSphere screen is visible and the anesthesiologist and PACU personal are instructed to follow the algorithm (chapter 4) in case of a HPI >85%. The purpose of the alarm at 85% and the presented algorithm is to prevent hypotension. If hypotension occurs, it should be treated as according to the standard of care.
  Interventions: Device: HPI (using HemoSphere) - guided algorithm
- Control group (Other): Patients in the control group are connected to the HemoSphere monitor to evaluate the TWA of hypotension in this group. The screen is not visible to the anesthesiologist or PACU personal and the alarm is set silent. It will be explained to the anesthesiologist and PACU personal that the patients are included to this study and that a blood pressure with a MAP of 65 mmHg should be monitored.
  Interventions: Device: Treatment of hypotension following standard of care

INTERVENTIONS:
Device: HPI (using HemoSphere) - guided algorithm — Treatment of hypotension guided by the hypotension prediction index. Patients will receive treatment following the predetermined HPI-algorithm when the HPI exceeds 85%.
  Arms: HPI-intervention algorithm
Device: Treatment of hypotension following standard of care — Patients receive standard of care treatment for hypotension, with a goal-mean arterial pressure (MAP) of 65mmHg.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate if the use of the hypotension prediction index during the perioperative period leads to a decrease in hypotension both during and after surgery (24 hrs) in adults undergoing major abdominal surgery. The main question this trial aims to answer is:

• Does the use of the hypertension prediction index (HPI) decrease hypotension during surgery and in the post-operative period?

During and after their surgery, participants in the intervention group will be treated according to the HPI-algorithm.

Participants in the control group will be treated following the standard of care.

DETAILED DESCRIPTION:
Rationale: Hypotension during and after surgery is associated with serious complications. Using a machine learning algorithm, hypotension can be accurately predicted. Edwards Lifesciences developed this algorithm, called "Hypotension Prediction Index" and integrated this in their hemodynamical monitors. Recent studies have shown a decrease in intraoperative hypotension when using the hypotension prediction index.

Objective: To investigate if the use of the hypotension prediction index during the perioperative period leads to a decrease in hypotension (time weighted average) both during and after surgery (24 hrs).

Intervention: Patients in the intervention group will be treated using the hypotension prediction index algorithm to prevent hypotension. In case of actual hypotension the treatment thereof is at the discretion of the anaesthesiologist.

Main study parameters/endpoints: The decrease in time weighted average of hypotension in the peri- and post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Patients planned to undergo laparotomy surgery
* Patients that will receive an invasive arterial catheter as part of their procedure
* Patients that are planned to go to the post anaesthetic care unit (PACU) post-operatively

Exclusion Criteria:

* Patients with known arrythmias
* Patients with known severe heart valve disease
* Patients with the need for dialysis
* Clamping of the aorta or Pringle's manoeuvre during surgery
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-22 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Time Weighted Average of hypotension | During the accumulative duration of surgery and PACU admission
  Time Weighted Average (TWA) is measured as (depth of hypotension in mmHg below a MAP op 65mmHg x time in minutes spent below a MAP of 65mmHg) ÷ total duration of surgery/PACU admission in minutes)

SECONDARY OUTCOMES:
Frequency and duration of hypotension | During surgery and in the 24 hours following surgery
  Defined as MAP<65mmHg for at least 1 minute
Frequency and duration of hypertension | During surgery and in the 24 hours following surgery
  Defined as MAP>100mmHg for at least 1 minute
Total amount of administered fluids | During surgery and in the 24 hours following surgery
  Total amount of administered fluids (absolute, ml/kg/min, input/output ratio)
Total administration of vasopressors | During surgery and in the 24 hours following surgery
  Total administration of vasopressors (mcg/kg/min)
Total administration of inotropy | During surgery and in the 24 hours following surgery
  Total administration of inotropy (mcg/kg/min)
Eligibility for discharge to the ward on the day after surgery | During morning rounds the day after surgery (approximately at 10.00hours)
  Eligibility defined as yes or no
Lactate | "at the start of surgery", "at PACU admission", "day after surgery at 06.00hours"
  Lactate level as measured in arterial blood gas
Glomerular filtration rate | "at the start of surgery", "at PACU admission", "day after surgery at 06.00hours"
  Glomerular filtration rate as measured in arterial blood gas
Number and type of complications in the first 30 days after surgery | 30 days after surgery
  Number and type of complications in the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Van Eijk, Principal Investigator — Coordinating Investigator

IPD SHARING:
Plan to Share IPD: No